CLINICAL TRIAL: NCT04659525
Title: Phase IV Study for Efficacy and Safety of Evolocumab Added to Ezetimibe (Standard of Care) in High Cardiovascular Risk Haemodialized Statin Intolerant Patients With Hypercholesterolemia
Brief Title: Evolocumab Plus Ezetimibe in Haemodialized Statin-intolerant Patients With Hypercholesterolemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Policlinico Casilino ASL RMB (Other)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Leonardo Calò, MD, Head of Cardiology Department, Policlinico Casilino ASL RMB
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Evolocumab02
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Hypercholesterolemia; CKD Stage 5; Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: Hypercholesterolemia; Chronic Dialysis; Statin intollerant patients; LDL reduction; Cardiovascular risk
MeSH Terms: conditions — Hypercholesterolemia; Renal Insufficiency, Chronic | interventions — evolocumab; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evolocumab + Ezetimibe (Experimental): Patients in this arm will receive subcutaneous evolocumab 140 mg every two weeks plus ezetimibe 10 mg per os daily for 24 weeks
  Interventions: Drug: Evolocumab; Drug: Ezetimibe
- Placebo + Ezetimibe (Placebo Comparator): Patients in this arm will receive subcutaneous placebo every two weeks plus ezetimibe 10 mg per os daily for 24 weeks
  Interventions: Drug: Ezetimibe; Drug: Placebo

INTERVENTIONS:
Drug: Evolocumab — In the intervention arm evolocumab 140 mg subcutaneous every 2 weeks will be administered for 24 weeks to high cardiovascular risk haemodialized statin intolerant patients with hypercholesterolemia
  Arms: Evolocumab + Ezetimibe
Drug: Ezetimibe — Ezetimibe 10 mg daily will be administered for 24 weeks to high cardiovascular risk haemodialized statin intolerant patients with hypercholesterolemia in both the placebo arm (plus placebo) and in the intervention arm (plus evolocumab)
Drug: Placebo — In the placebo arm placebo subcutaneous every 2 weeks will be administered for 24 weeks to high cardiovascular risk haemodialized statin intolerant patients with hypercholesterolemia
  Arms: Placebo + Ezetimibe

SUMMARY:
Evolocumab is a monoclonal antibody that inhibits proprotein convertase subtilisin-kexin type 9 (PCSK9) and lowers low-density lipoprotein (LDL) cholesterol, reducing in turn the risk of cardiovascular events. Whether evolcumab is effective in haemodialized patients is uncertain. The investigators will conduct a randomized, double-blind, placebo-controlled trial to assess the feasibility, safety, and LDL-C-lowering efficacy of evolocumab in high cardiovascular risk haemodialized statin intolerant patients with hypercholesterolemia. Patients will be randomly assigned to receive evolocumab (140 mg subcutaneous every 2 weeks + ezetimibe 10 mg per os daily) or matching placebo (subcutaneous every 2 weeks + ezetimibe 10 mg per os daily) for 24 weeks. The primary efficacy end point will be the proportion of patients that will reduce LDL-C < 55 mg/dL in the evolocumab group compared to placebo at 24 weeks. The key secondary efficacy end points will be: the reduction of LDL-C from baseline at 4, 6 and 12 weeks; the reduction of HDL-C, non-HDL cholesterol and triglycerides from baseline at 24 weeks. Every adverse event (serious and non-serious) correlated to drug infusion will be recorded (safety end-point).

ELIGIBILITY:
Inclusion Criteria:

* high cardiovascular risk defined as patients with: Documented cardiovascular disease (CVD), clinical or unequivocal on imaging. Documented clinical CVD includes previous acute myocardial infarction, coronary revascularization and other arterial revascularization procedures, stroke and TIA, aortic aneurysm and PAD. Unequivocally documented CVD on imaging includes plaque on coronary angiography or carotid ultrasound; DM with target organ damage or with a major risk factor such as smoking or marked hypercholesterolaemia or marked hypertension.
* History of statin intolerance, demonstrated by: trial of ≥2 statins with intolerance of any dose or to increase statin dose above the total maximum doses because of intolerable: Myopathy or myalgia (muscle pain, ache, or weakness without CK elevation), or Myositis (muscle symptoms with increased CK levels), or Rhabdomyolysis (muscle symptoms with marked CK elevation) and Resolution or improvement of symptoms when the statin dose was decreased or discontinued
* patients with LDL-C >55 mg/dL
* end-stage renal disease on chronic hemodialysis
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* secondary hypercholesterolemia (i.e. hypothyroidism, Primary biliary cholangitis, etc)
* Use of drugs or dietary supplements that can impact on cholesterol value (i.e. progestinic, red yeast rice, niacin >200 mg/d, lipid-regulating drugs - eg, ﬁbrates or derivatives, ezetimibe, bile-acid sequestrants, stanols, or stanol esters - )
* Previous treatment with evolocumab or any other anti-PCSK9 therapy
* Inability to provide informed consent or to attend follow-up visits
* Unreliability as a study participant based on judgment of investigator's knowledge of the subject (eg, alcohol or other drug abuse, inability or unwillingness to adhere to the protocol, psychosis)
* Current enrollment in another investigational device or drug study or <30 d since ending another investigational device or drug study
* serum triglycerides level > 400 mg/dL at baseline
* Pregnancy, breastfeeding, or inadequate birth control in premenopausal female subjects
* Laboratory values at screening CK >3 × ULN; AST or ALT >2 × ULN

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
LDL cholesterol change dichotomic | 24 weeks
  proportion of patients that achieve an LDL cholesterol level < 55 mg/dL

SECONDARY OUTCOMES:
LDL cholesterol change time-points | 4 weeks, 12 weeks, 24 weeks
  change in LDL cholesterol levels from baseline
HDL cholesterol change | 24 weeks
  change in HDL cholesterol levels from baseline
non-HDL cholesterol change | 24 weeks
  change in non-HDL cholesterol levels from baseline
Triglycerides change | 24 weeks
  change in triglycerides levels from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Casilino, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mach F, Baigent C, Catapano AL, Koskinas KC, Casula M, Badimon L, Chapman MJ, De Backer GG, Delgado V, Ference BA, Graham IM, Halliday A, Landmesser U, Mihaylova B, Pedersen TR, Riccardi G, Richter DJ, Sabatine MS, Taskinen MR, Tokgozoglu L, Wiklund O; ESC Scientific Document Group. 2019 ESC/EAS Guidelines for the management of dyslipidaemias: lipid modification to reduce cardiovascular risk. Eur Heart J. 2020 Jan 1;41(1):111-188. doi: 10.1093/eurheartj/ehz455. No abstract available. PMID 31504418
- [Background] Wanner C, Krane V, Marz W, Olschewski M, Mann JF, Ruf G, Ritz E; German Diabetes and Dialysis Study Investigators. Atorvastatin in patients with type 2 diabetes mellitus undergoing hemodialysis. N Engl J Med. 2005 Jul 21;353(3):238-48. doi: 10.1056/NEJMoa043545. PMID 16034009
- [Background] Fellstrom BC, Jardine AG, Schmieder RE, Holdaas H, Bannister K, Beutler J, Chae DW, Chevaile A, Cobbe SM, Gronhagen-Riska C, De Lima JJ, Lins R, Mayer G, McMahon AW, Parving HH, Remuzzi G, Samuelsson O, Sonkodi S, Sci D, Suleymanlar G, Tsakiris D, Tesar V, Todorov V, Wiecek A, Wuthrich RP, Gottlow M, Johnsson E, Zannad F; AURORA Study Group. Rosuvastatin and cardiovascular events in patients undergoing hemodialysis. N Engl J Med. 2009 Apr 2;360(14):1395-407. doi: 10.1056/NEJMoa0810177. Epub 2009 Mar 30. PMID 19332456
- [Background] Baigent C, Landray MJ, Reith C, Emberson J, Wheeler DC, Tomson C, Wanner C, Krane V, Cass A, Craig J, Neal B, Jiang L, Hooi LS, Levin A, Agodoa L, Gaziano M, Kasiske B, Walker R, Massy ZA, Feldt-Rasmussen B, Krairittichai U, Ophascharoensuk V, Fellstrom B, Holdaas H, Tesar V, Wiecek A, Grobbee D, de Zeeuw D, Gronhagen-Riska C, Dasgupta T, Lewis D, Herrington W, Mafham M, Majoni W, Wallendszus K, Grimm R, Pedersen T, Tobert J, Armitage J, Baxter A, Bray C, Chen Y, Chen Z, Hill M, Knott C, Parish S, Simpson D, Sleight P, Young A, Collins R; SHARP Investigators. The effects of lowering LDL cholesterol with simvastatin plus ezetimibe in patients with chronic kidney disease (Study of Heart and Renal Protection): a randomised placebo-controlled trial. Lancet. 2011 Jun 25;377(9784):2181-92. doi: 10.1016/S0140-6736(11)60739-3. Epub 2011 Jun 12. PMID 21663949
- [Background] Stroes E, Colquhoun D, Sullivan D, Civeira F, Rosenson RS, Watts GF, Bruckert E, Cho L, Dent R, Knusel B, Xue A, Scott R, Wasserman SM, Rocco M; GAUSS-2 Investigators. Anti-PCSK9 antibody effectively lowers cholesterol in patients with statin intolerance: the GAUSS-2 randomized, placebo-controlled phase 3 clinical trial of evolocumab. J Am Coll Cardiol. 2014 Jun 17;63(23):2541-2548. doi: 10.1016/j.jacc.2014.03.019. Epub 2014 Mar 30. PMID 24694531
- [Background] Schwartz GG, Steg PG, Szarek M, Bhatt DL, Bittner VA, Diaz R, Edelberg JM, Goodman SG, Hanotin C, Harrington RA, Jukema JW, Lecorps G, Mahaffey KW, Moryusef A, Pordy R, Quintero K, Roe MT, Sasiela WJ, Tamby JF, Tricoci P, White HD, Zeiher AM; ODYSSEY OUTCOMES Committees and Investigators. Alirocumab and Cardiovascular Outcomes after Acute Coronary Syndrome. N Engl J Med. 2018 Nov 29;379(22):2097-2107. doi: 10.1056/NEJMoa1801174. Epub 2018 Nov 7. PMID 30403574
- [Background] Sabatine MS, Giugliano RP, Keech AC, Honarpour N, Wiviott SD, Murphy SA, Kuder JF, Wang H, Liu T, Wasserman SM, Sever PS, Pedersen TR; FOURIER Steering Committee and Investigators. Evolocumab and Clinical Outcomes in Patients with Cardiovascular Disease. N Engl J Med. 2017 May 4;376(18):1713-1722. doi: 10.1056/NEJMoa1615664. Epub 2017 Mar 17. PMID 28304224